CLINICAL TRIAL: NCT05552027
Title: Sensor Network With Active Instructional Content to Prevent Child Safety Seat Misuse
Brief Title: Minnesota HealthSolutions Cellular Car Seat Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minnesota HealthSolutions (Industry)
Collaborators: Children's Hospital of Philadelphia (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sara Seifert, MPH, Minnesota HealthSolutions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20-017790
Record Dates: First submitted 2022-08-05; First posted 2022-09-23 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Child Safety Seat Harness Tension

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial with 2 arms (intervention and control). The intervention group will participate in a series of three safety seat misuse scenarios with the CCS system enabled, and participants in the control group will participate in the same series of three safety seat misuse scenarios without the CCS system. Misuse scenarios include insecure attachment of the seat to the vehicle, incorrect harness straps, and improper orientation of the safety seat. In each scenario, participants will be asked to identify and correct each error. Each participant will be randomly assigned to either the control or intervention group. Each participant will receive the same scenarios in the same order.
Who Masked: Participant
Masking Description: Participants will be randomly assigned to the intervention group or control group upon arrival at the study visit. Assignment status will not be concealed from the research assistants enrolling the participant, the participants themselves, or the rest of the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will harness the car seat in 3 separate scenarios with the sensor system enabled to provide feedback.
  Interventions: Device: CCS System- Prototype
- Control (Other): Participants will harness the car seat in 3 separate scenarios with the sensor system disabled in order to not provide feedback.
  Interventions: Device: CCS System- Control

INTERVENTIONS:
Device: CCS System- Prototype — Participants will be exposed to each of the 3 scenarios with the sensor system enabled (with feedback)
  Arms: Intervention
Device: CCS System- Control — The participants will be exposed to each of the 3 scenarios with the system disabled (no feedback).
  Arms: Control

SUMMARY:
The objective of the study is to evaluate an innovative child safety seat user engagement system (CCS system) designed to actively educate, instruct, and alarm caregivers with information associated with automatically-sensed safety seat misuses/errors via a smartphone application.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate whether child safety seat users correct more critical misuse errors in child safety seat usage with the seat with the CCS system than the same seat with no sensor system. The CCS system will provide ongoing, tailored support to users at the time of an error. Videos will be available to users via a smartphone and provide short "how to" instructions that demonstrate how to correctly perform each safety seat behavior (e.g., tighten harness straps) and how to avoid common mistakes. The overall goal of the CCS system is to prevent child safety seat critical misuses and reduce deaths and injuries in children riding in motor vehicles. In the proposed study, adult participants will be asked to attend one in-person study visit and complete three (3) scenarios in which they will be asked to identify and correct errors in child safety seat use. Participants will be randomized to either the intervention group which will use the CCS system during each scenario or the control group which will not use the CCS system during each scenario.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females ages 18-75 years
* Has harnessed/fastened a child into a car seat in the last five (5) years
* Has a valid driver's license

Exclusion Criteria:

* Non-fluency in written and/or spoken English
* Participant cannot install a safety seat due to a physical or health limitation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Seifert, MPH, Principal Investigator — Minnesota HealthSolutions
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and study documents will be shared with Minnesota HealthSolutions (the sponsor). No identifiable data will be used for future study without first obtaining Institutional Review Board (IRB) approval. The investigator will obtain a data use agreement between the provider (the PI) of the data and any recipient researchers (including others at CHOP) before sharing a limited dataset (PHI limited to dates and zip codes).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study will comply with CHOP's data retention policy (A-3-9). All study data will be maintained for at least 6 years following study completion. There is no set timeline for the destruction of the study's de-identified data
Access Criteria: IRB approval, data use agreement

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Ten leading causes of unintentional injury deaths, United States, 2016, all races, both sexes. https://webappa.cdc.gov/cgi-bin/broker.exe. Published 2016.
- [Background] Centers for Disease Control and Prevention. Fatal Injury Data. https://www.cdc.gov/injury/wisqars/fatal.html. Accessed January 5, 2019.
- [Background] National Highway Traffic Safety Administration. Traffic Safety Facts 2008 Data: Young Drivers. Vol 2010. Washington, DC: US Department of Transportation; 2008. doi:DOT HS 811 169
- [Background] National SAFE KIDS Campaign and NHTSA Child Passenger Safety Technician Program Participant Manual. :C-4.
- [Background] Li HR, Pickrell TM, KC S. The 2015 National Survey of the Use of Booster Seats. Washington, DC; 2016. www.ntis.gov.
- [Background] Greenwell NK. Results of the National Child Restraint Use Special Study. Washington, DC; 2015. www.ntis.gov.
- [Background] Durbin DR, Elliott MR, Winston FK. Belt-positioning booster seats and reduction in risk of injury among children in vehicle crashes. JAMA. 2003 Jun 4;289(21):2835-40. doi: 10.1001/jama.289.21.2835. PMID 12783914
- [Background] Arbogast KB, Durbin DR, Cornejo RA, Kallan MJ, Winston FK. An evaluation of the effectiveness of forward facing child restraint systems. Accid Anal Prev. 2004 Jul;36(4):585-9. doi: 10.1016/S0001-4575(03)00065-4. PMID 15094411
- [Background] Brown J, Bilston L, McCaskill M. Injury implications of inappropriate use of adult seatbelt systems for children aged 2-8. Australas Road Res Polic Educ Conf. 2003;7(2):81-87.
- [Background] Brown J, McCaskill ME, Henderson M, Bilston LE. Serious injury is associated with suboptimal restraint use in child motor vehicle occupants. J Paediatr Child Health. 2006 Jun;42(6):345-9. doi: 10.1111/j.1440-1754.2006.00870.x. PMID 16737475
- [Background] Lutz N, Arbogast KB, Cornejo RA, Winston FK, Durbin DR, Nance ML. Suboptimal restraint affects the pattern of abdominal injuries in children involved in motor vehicle crashes. J Pediatr Surg. 2003 Jun;38(6):919-23. doi: 10.1016/s0022-3468(03)00124-6. PMID 12778394
- [Background] Valent F, McGwin G Jr, Hardin W, Johnston C, Rue LW 3rd. Restraint use and injury patterns among children involved in motor vehicle collisions. J Trauma. 2002 Apr;52(4):745-51. doi: 10.1097/00005373-200204000-00023. PMID 11956394
- [Background] Weinstein EB, Sweeney MM, Garber M, Eastwood MD, Osterman JG, Roberts JV. The Effect of Size Appropriate and Proper Restraint Use on Injury Severity of Children. In: 2nd Child Occupant Protection Symposium. Society of Automotive Engineers (SAE); 1997:181-186.
- [Background] Winston FK, Durbin DR, Kallan MJ, Moll EK. The danger of premature graduation to seat belts for young children. Pediatrics. 2000 Jun;105(6):1179-83. doi: 10.1542/peds.105.6.1179. PMID 10835054
- [Background] Decina LE, Lococo KH. Misuse of child restraints. 2004. http://icsw.nhtsa.gov/people/injury/research/misuse/images/misusescreen.pdf.
- [Background] Klinich KD, Manary MA, Flannagan CAC, et al. Labels, Instructions, and Features of Convertible Child Restraint Systems (CRS): Evaluating Their Effects on CRS Installation Errors. Washington, DC; 2010.
- [Background] Wegner MV, Girasek DC. How readable are child safety seat installation instructions? Pediatrics. 2003 Mar;111(3):588-91. doi: 10.1542/peds.111.3.588. PMID 12612241
- [Background] Doak CC, Doak LG, Root JH. Teaching Patients with Low Literacy Skills. 2nd ed. Philadelphia: JB Lippincott Co.; 1996.
- [Background] Participants Central. Prevent child heatsroke in cars. http://www.safercar.gov/participants/InandAroundtheCar/heatstroke.htm. Accessed December 7, 2016.
- [Background] Singh S, Stern S, Subramanian R. Not-in-Traffic Surveillance: Non-Crash Fatalities and Injuries.; 2015.
- [Background] Rudd R, Prasad A, Weston D, Wietholter K. Functional Assessment of Unattended Child Reminder Systems. Washington, DC; 2015.
- [Background] Null J. Heatsroke deaths of children in vehicles. https://noheatstroke.org/index.htm. Accessed January 5, 2019.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 46 | 46
Completed | 46 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 46 | 92
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [31 to 59] | 36 [24 to 44] | 36 [24 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 44 | 41 | 85
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 33 | 23 | 56
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Installation Errors
Description: For each misuse scenario participants will be asked to correct the error in the seat installation or the harness tension. Convertible seats will be used for this phase. For each scenario, we will use a huggable images test doll (age and weight of the doll will be indicated to participants). Study team will record seat direction (forward vs rear facing), harness tension (newtons), insecure attachment of the seat to the vehicle (yes/no).
Time Frame: Once during the only study visit: up to 30 mins
Population: Participants in the intervention group were given a study phone and asked to use the CCS smartphone app to complete the scenarios, while the control group was given only the paper manual that came with the safety seat. The misuse scenarios included A) a full safety seat installation with the convertible seat beginning on the floor, B) loose harness straps, and C) loose attachment to the vehicle seat at the base.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention - Scenario A: Sensor system enabled to provide feedback. Full seat installation.
- Control - Scenario A: Sensor system disabled in order to not provide feedback. Full seat Installation.
- Intervention - Scenario B: Sensor enabled to provide feedback. Harness straps left loose.
- Control - Scenario B: Sensor system disabled in order to not provide feedback. Harness straps left loose.
- Intervention - Scenario C: Sensor system enabled. Carseat left loose at the base.
- Control - Scenario C: Sensor system disable to not provide feedback. Carseat left loose at the base.
Arm/Group | Intervention - Scenario A | Control - Scenario A | Intervention - Scenario B | Control - Scenario B | Intervention - Scenario C | Control - Scenario C
Number analyzed (Participants) | 46 | 46 | 46 | 46 | 46 | 46
Participants | 21 | 41 | 17 | 32 | 18 | 33
Statistical Analysis 1: Comparison: Intervention - Scenario A vs Control - Scenario A; Test type: Superiority; p < .001, Chi-squared — At the completion of scenario A (a full child safety seat installation), the participants using the CCS app had significantly fewer errors present compared to the control group
Statistical Analysis 2: Comparison: Intervention - Scenario B vs Control - Scenario B; Test type: Superiority; p < .01, Chi-squared — At the end of scenario B (loose harness straps), participants using the CCS app had significantly fewer errors present compared to the control group
Statistical Analysis 3: Comparison: Intervention - Scenario C vs Control - Scenario C; Test type: Superiority; p < .01, Chi-squared — At the end of scenario C (loose attachment at the base), like the other two scenarios, participants using the CCS app had significantly fewer errors present compared to the control group

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- Intervention: CCS System Enabled. There are no adverse events to record for this study group.
- Control: CCS System Disabled. There are no adverse events to record for this study group.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT05552027/Prot_000.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT05552027/ICF_001.pdf